CLINICAL TRIAL: NCT02174861
Title: An Open-label Extension (OLE) Study to Assess the Long-term Safety and Efficacy of AMG 334
Brief Title: A Study to Assess the Long-term Safety and Efficacy of Erenumab (AMG 334) in Chronic Migraine Prevention.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130255; 2013-005311-27 (EudraCT Number)
Record Dates: First submitted 2014-05-28; First posted 2014-06-26 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Treatment for Prevention of Chronic Migraine
Keywords: Chronic Migraine
MeSH Terms: interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erenumab (Experimental): Participants received erenumab 70 mg once a month (QM) or 140 mg QM by subcutaneous injection for up to 52 weeks.
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Erenumab — Administered by subcutaneous injection once a month
  Other Names: AMG 334; Aimovig™

SUMMARY:
To assess the long-term safety and efficacy of erenumab.

DETAILED DESCRIPTION:
This was a multicenter, 52-week, open-label study designed to assess the long-term safety and efficacy of erenumab in adults with chronic migraine. Participants who completed the 12-week double-blind treatment of the parent Study 20120295 (NCT02066415) and met all Study 20130255 eligibility criteria were eligible for enrollment into this study. Enrollment occurred within 14 days after the parent study's week 12 visit.

The initial dose used in the study was erenumab 70 mg every month (QM). The protocol was subsequently amended to increase the dose to erenumab 140 mg QM (Protocol Amendment 2). Participants who had already completed the week 28 visit (ie, midpoint of the study) at the time of Protocol Amendment 2 continued to receive open-label erenumab 70 mg QM for the remainder of the study. Participants who enrolled but had not completed the week 28 visit at the time of Protocol Amendment 2 increased the open-label erenumab dose from 70 mg QM to 140 mg QM at the next visit. All participants who enrolled after Protocol Amendment 2 received open-label erenumab 140 mg QM throughout the study.

Participants may elect to participate in a separate clinical home use (CHU) substudy to assess subjects' ability to self-administer 140 mg of erenumab for in-home use using either two prefilled syringes (PFS) or two prefilled autoinjector/pens (AI/pens). Enrollment in the 12-week substudy occurred at either week 12 or week 40 of study 20130255. Participants were randomized to self-administer erenumab using either the PFS or AI/pen on CHU days 29 and 57 at home.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent prior to initiation of any study-specific activities/procedures
2. Completed the 12-week study visit and did not end IP early during the double-blind treatment period of the AMG 334 20120295 (NCT02066415) parent study, and is appropriate for continued treatment.

Exclusion Criteria:

1. Development of any unstable or clinically significant medical condition, laboratory or electrocardiogram (ECG) abnormality following randomization into the parent study, that in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
2. Systolic blood pressure (BP) 160 mm Hg and/or diastolic BP 100 mm Hg or greater at screening/Day 1.
3. Subject who used excluded concomitant medications between week 8 and week 12 of the parent study

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (59):
- United States (28):
  - Research Site, Newport Beach, California
  - Research Site, Palo Alto, California
  - Research Site, Santa Monica, California
  - Research Site, Sherman Oaks, California
  - Research Site, Stamford, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Beach Gardens, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Indianapolis, Indiana
  - Research Site, Pikesville, Maryland
  - Research Site, Watertown, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Reno, Nevada
  - Research Site, Amherst, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Virginia Beach, Virginia
  - Research Site, Seattle, Washington
- Canada (2):
  - Research Site, Calgary, Alberta
  - Research Site, Montreal, Quebec
- Czechia (2):
  - Research Site, Brno
  - Research Site, Prague
- Research Site, Glostrup Municipality, Denmark
- Finland (4):
  - Research Site, Helsinki
  - Research Site, Oulu
  - Research Site, Tampere
  - Research Site, Turku
- Germany (5):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Kiel
- Norway (4):
  - Research Site, Ålesund
  - Research Site, Lillehammer
  - Research Site, Sandvika
  - Research Site, Stavanger
- Poland (6):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Świdnik
  - Research Site, Warsaw
- Sweden (3):
  - Research Site, Falköping
  - Research Site, Stockholm
  - Research Site, Vällingby
- United Kingdom (4):
  - Research Site, Glasgow
  - Research Site, Hull
  - Research Site, London
  - Research Site, Stoke-on-Trent

REFERENCES:
- [Background] Zhou Y, Zhang F, Starcevic Manning M, Hu Z, Hsu CP, Chen PW, Peng C, Loop B, Mytych DT, Paiva da Silva Lima G. Immunogenicity of erenumab: A pooled analysis of six placebo-controlled trials with long-term extensions. Cephalalgia. 2022 Jul;42(8):749-760. doi: 10.1177/03331024221075621. Epub 2022 Mar 10. PMID 35272533
- [Background] Ashina M, Kudrow D, Reuter U, Dolezil D, Silberstein S, Tepper SJ, Xue F, Picard H, Zhang F, Wang A, Zhou Y, Hong F, Klatt J, Mikol DD. Long-term tolerability and nonvascular safety of erenumab, a novel calcitonin gene-related peptide receptor antagonist for prevention of migraine: A pooled analysis of four placebo-controlled trials with long-term extensions. Cephalalgia. 2019 Dec;39(14):1798-1808. doi: 10.1177/0333102419888222. Epub 2019 Nov 10. PMID 31707815
- [Derived] Ashina M, Goadsby PJ, Dodick DW, Tepper SJ, Xue F, Zhang F, Brennan F, Paiva da Silva Lima G. Assessment of Erenumab Safety and Efficacy in Patients With Migraine With and Without Aura: A Secondary Analysis of Randomized Clinical Trials. JAMA Neurol. 2022 Feb 1;79(2):159-168. doi: 10.1001/jamaneurol.2021.4678. PMID 34928306
- [Derived] Tepper SJ, Ashina M, Reuter U, Hallstrom Y, Broessner G, Bonner JH, Picard H, Cheng S, Chou DE, Zhang F, Klatt J, Mikol DD. Reduction in acute migraine-specific and non-specific medication use in patients treated with erenumab: post-hoc analyses of episodic and chronic migraine clinical trials. J Headache Pain. 2021 Jul 23;22(1):81. doi: 10.1186/s10194-021-01292-w. PMID 34301173
- [Derived] Tepper SJ, Ashina M, Reuter U, Brandes JL, Dolezil D, Silberstein SD, Winner P, Zhang F, Cheng S, Mikol DD. Long-term safety and efficacy of erenumab in patients with chronic migraine: Results from a 52-week, open-label extension study. Cephalalgia. 2020 May;40(6):543-553. doi: 10.1177/0333102420912726. Epub 2020 Mar 26. PMID 32216456
- [Derived] Kudrow D, Pascual J, Winner PK, Dodick DW, Tepper SJ, Reuter U, Hong F, Klatt J, Zhang F, Cheng S, Picard H, Eisele O, Wang J, Latham JN, Mikol DD. Vascular safety of erenumab for migraine prevention. Neurology. 2020 Feb 4;94(5):e497-e510. doi: 10.1212/WNL.0000000000008743. Epub 2019 Dec 18. PMID 31852816
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 64 centers across North America and Europe from 30 June 2014 to 4 March 2016. Participants who completed the 12-week double-blind treatment of the parent Study 20120295 (NCT02066415) and met all Study 20130255 eligibility criteria were eligible for enrollment into this study.
Pre-assignment Details: Participants at sites in the United States, Sweden, and Germany had the option of enrolling in the Clinical Home Use (CHU) Substudy to assess their ability to self-administer 140 mg erenumab for in-home use. Participants in the substudy were randomized 1:1 to self-administer erenumab using either a prefilled syringe or autoinjector/pen.
Groups:
- Erenumab: Participants received erenumab 70 mg once a month (QM) and/or 140 mg QM by subcutaneous injection for up to 52 weeks.
  Participants who enrolled prior to amendment 2 received erenumab 70 mg once a month (QM). Participants who had not completed the week 28 visit at the time of amendment 2 had their dose increased to 140 mg QM at their next visit whereas participants who had already completed the week 28 visit remained on erenumab 70 mg QM. Participants who enrolled after amendment 2 received erenumab 140 mg QM for the duration of the study.
Period: Overall Study
Arm/Group | Erenumab
Started | 609
Enrolled in CHU Substudy | 53
Completed | 451
Not Completed | 158
Not completed — Decision by sponsor | 8
Not completed — Withdrawal by Subject | 124
Not completed — Lost to Follow-up | 26

BASELINE CHARACTERISTICS:
Arm/Group | Erenumab
Number analyzed (Participants) | 609
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (11.3)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 608
  65 - 74 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 509
  Male | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 584
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Black or African American | 25
  Native Hawaiian or Other Pacific Islander | 0
  White | 574
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were graded for severity using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, where Grade 1 = mild AE, asymptomatic or mild symptoms; Grade 2 = Moderate AE; Grade 3 = Severe or medically significant but not immediately life-threatening; Grade 4 = Life-threatening consequences; urgent intervention indicated; Grade 5 = Death related to AE.
Time Frame: From first dose of erenumab in extension study 20130255 to the end of the 12-week safety follow-up period (up to 64 weeks).
Population: All enrolled participants who received at least 1 dose of erenumab
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab
Number analyzed (Participants) | 609
Participants
  Any adverse event | 398
  Adverse event grade ≥ 2 | 302
  Adverse event grade ≥ 3 | 34
  Adverse event grade ≥ 4 | 0
  Treatment-related adverse events | 114
  Serious adverse events | 24
  AE leading to discontinuation of erenumab | 16
  Fatal adverse events | 0

2. Primary Outcome: CHU Substudy: Number of Participants Able to Administer a Full Dose of Erenumab in Home-use
Description: At the CHU substudy day 28 and day 56 visits, the site provided erenumab 140 mg to participants to self-administer at home on the following day. Study site staff then called the participants and asked if they administered a full, partial, or no dose of erenumab. A full dose was defined when the entire volume of both prefilled syringes or autoinjector/pens were injected.
Time Frame: Day 29 (week 4) and day 57 (week 8) of the substudy
Population: All randomized participants who received at least 1 dose of erenumab in the CHU substudy.
Measure: Count of Participants; unit: Participants
Groups:
- Erenumab 140 mg PFS: Participants in the CHU substudy self-administered erenumab 140 mg on days 29 and 57 by subcutaneous injection using a prefilled syringe (PFS).
- Erenumab 140 mg AI/Pen: Participants in the CHU substudy self-administered erenumab 140 mg on days 29 and 57 by subcutaneous injection using a autoinjector/pen (AI/Pen).
Arm/Group | Erenumab 140 mg PFS | Erenumab 140 mg AI/Pen
Number analyzed (Participants) | 27 | 26
Participants
  Week 4 | 25 | 26
  Week 8 | 25 | 25

3. Secondary Outcome: Change From Study 20120295 Baseline in Monthly Migraine Days
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine with or without aura.
  The change from baseline in monthly migraine days was calculated as the number of migraine days during the 4 weeks prior to each study visit - the number of migraine days during the 4-week baseline phase.
Time Frame: 4-week baseline phase of Study 20120295 and the 4 weeks prior to the week 4, 8, 12, 24, 40, and 52 visits of Study 20130255
Population: Enrolled participants who received at least one dose of erenumab and had at least one change from baseline measurement in monthly migraine day in study 20130255. The number of participants analyzed includes participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: migraine days / month
Arm/Group | Erenumab
Number analyzed (Participants) | 605
migraine days / month
  Baseline | 18.11 (4.53)
  Change from baseline at week 4: number analyzed (Participants) | 561
  Change from baseline at week 4 | -6.72 (6.22)
  Change from baseline at week 8: number analyzed (Participants) | 574
  Change from baseline at week 8 | -7.38 (6.50)
  Change from baseline at week 12: number analyzed (Participants) | 560
  Change from baseline at week 12 | -7.63 (6.49)
  Change from baseline at week 24: number analyzed (Participants) | 481
  Change from baseline at week 24 | -8.36 (6.29)
  Change from baseline at week 40: number analyzed (Participants) | 430
  Change from baseline at week 40 | -8.72 (6.53)
  Change from baseline at week 52: number analyzed (Participants) | 383
  Change from baseline at week 52 | -9.29 (6.64)

4. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction in Monthly Migraine Days From Study 20120295 Baseline
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine without aura or a migraine with aura. Monthly migraine days were calculated as the number of migraine days in the 4-week baseline phase and during the 4 weeks prior to each study visit.
  At least a 50% reduction from baseline (of study 20120295) in monthly migraine days was determined if the change in monthly migraine days from the 4-week baseline phase to the 4 weeks prior to each study visit * 100 / baseline monthly migraine days was less than or equal to -50%.
Time Frame: 4-week baseline phase of Study 20120295 and the 4 weeks prior to the week 4, 8, 12, 24, 40 and 52 visits of Study 20130255
Population: Enrolled participants who received at least one dose of erenumab and had at least one change from baseline measurement in monthly migraine day in study 20130255. The analysis includes participants with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erenumab
Number analyzed (Participants) | 605
percentage of participants
  Week 4: number analyzed (Participants) | 561
  Week 4 | 39.2 [35.3 to 43.3]
  Week 8: number analyzed (Participants) | 574
  Week 8 | 45.6 [41.6 to 49.7]
  Week 12: number analyzed (Participants) | 560
  Week 12 | 45.7 [41.6 to 49.9]
  Week 24: number analyzed (Participants) | 481
  Week 24 | 53.6 [49.2 to 58.0]
  Week 40: number analyzed (Participants) | 430
  Week 40 | 55.6 [50.9 to 60.2]
  Week 52: number analyzed (Participants) | 383
  Week 52 | 59.0 [54.0 to 63.8]

5. Secondary Outcome: Change From Study 20120295 Baseline in Monthly Acute Migraine-Specific Medication Treatment Days
Description: Monthly acute migraine-specific medication treatment days is the number of days on which migraine specific medications were used between monthly doses of study drug. Migraine-specific medications includes two categories of medications: triptan-based migraine medications and ergotamine-based migraine medications.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: acute migraine treatment days / month
Arm/Group | Erenumab
Number analyzed (Participants) | 605
acute migraine treatment days / month
  Baseline | 9.53 (7.26)
  Change from baseline at Week 4: number analyzed (Participants) | 561
  Change from baseline at Week 4 | -3.59 (4.62)
  Change from baseline at Week 8: number analyzed (Participants) | 574
  Change from baseline at Week 8 | -4.01 (4.96)
  Change from baseline at Week 12: number analyzed (Participants) | 560
  Change from baseline at Week 12 | -3.96 (5.03)
  Change from baseline at Week 24: number analyzed (Participants) | 481
  Change from baseline at Week 24 | -4.39 (4.99)
  Change from baseline at Week 40: number analyzed (Participants) | 430
  Change from baseline at Week 40 | -4.58 (5.00)
  Change from baseline at Week 52: number analyzed (Participants) | 383
  Change from baseline at Week 52 | -4.97 (5.33)

6. Secondary Outcome: Change From Study 20120295 Baseline in Cumulative Monthly Headache Hours
Description: The cumulative duration of any qualified headache between monthly doses of study drug regardless of acute treatment use.
  A qualified headache was defined as follows:
  * a qualified migraine headache (including an aura-only event that is treated with acute migraine-specific medication), or
  * a qualified non-migraine headache, which is a headache that lasted continuously for ≥ 4 hours and was not a qualified migraine headache, or
  * a headache of any duration for which acute headache treatment was administered.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours / month
Arm/Group | Erenumab
Number analyzed (Participants) | 605
hours / month
  Baseline | 226.84 (125.54)
  Change from baseline at week 4: number analyzed (Participants) | 561
  Change from baseline at week 4 | -79.38 (107.56)
  Change from baseline at week 8: number analyzed (Participants) | 574
  Change from baseline at week 8 | -85.24 (110.24)
  Change from Baseline at week 12: number analyzed (Participants) | 560
  Change from Baseline at week 12 | -89.30 (111.47)
  Change from Baseline at week 24: number analyzed (Participants) | 481
  Change from Baseline at week 24 | -100.41 (112.30)
  Change from Baseline at week 40: number analyzed (Participants) | 430
  Change from Baseline at week 40 | -101.07 (111.77)
  Change from Baseline at week 52: number analyzed (Participants) | 383
  Change from Baseline at week 52 | -107.44 (113.60)

7. Secondary Outcome: CHU Substudy: Number of Participants With Adverse Events
Description: Adverse events were graded for severity using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
  Injection site reactions were derived from a Medical Dictionary for Regulatory Activities (MedDRA) query using a list of pre-specified preferred terms.
  An adverse device effect (ADE) is any adverse event related to the use of a medical device.
Time Frame: From first dose of erenumab in the CHU substudy to 28 days after last dose of erenumab in the CHU substudy; up to 12 weeks.
Population: All randomized participants who received at least one dose of erenumab in the CHU substudy.
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab 140 mg PFS | Erenumab 140 mg AI/Pen
Number analyzed (Participants) | 27 | 26
Participants
  Any adverse event | 2 | 6
  Adverse event grade ≥ 2 | 1 | 4
  Adverse event grade ≥ 3 | 0 | 0
  Adverse event grade ≥ 4 | 0 | 0
  Serious adverse events | 0 | 0
  AE leading to discontinuation of erenumab | 0 | 0
  Fatal adverse events | 0 | 0
  Injection site reactions | 0 | 1
  Adverse device effects | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of erenumab in extension study 20130255 to the end of the 12-week safety follow-up period (up to 64 weeks).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Erenumab
All-Cause Mortality (participants affected / at risk) | 0/609
Serious Adverse Events (participants affected / at risk) | 24/609
Other Adverse Events (participants affected / at risk) | 162/609
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab (N=609)
Myocardial bridging (Congenital, familial and genetic disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
Alcoholic liver disease (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Post procedural oedema (Injury, poisoning and procedural complications) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Medication overuse headache (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 4
Presyncope (Nervous system disorders) | 1
Radicular syndrome (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Vestibular migraine (Nervous system disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab (N=609)
Sinusitis (Infections and infestations) | 44
Upper respiratory tract infection (Infections and infestations) | 45
Viral upper respiratory tract infection (Infections and infestations) | 96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/61/NCT02174861/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT02174861/SAP_001.pdf